CLINICAL TRIAL: NCT00342173
Title: Costa Rican Natural History Study of HPV and Cervical Neoplasia
Status: Terminated | Type: Observational
Why Stopped: classified by the IRB as non human subjects research
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 999999030; OH99-C-N030
Record Dates: First submitted 2006-06-19; First posted 2006-06-21 (Estimated); Last update posted 2020-03-16 (Actual); Status verified 2020-03

CONDITIONS: Cervical Neoplasia
Keywords: Cervix; Natural History; Neoplasia; HPV; Costa Rica
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Women in Costa Rica: Examining the natural history of HPV and cervical neoplasia in Costa Rican women.

SUMMARY:
A population-based study was initiated in Costa Rica in June 1993 to investigate the natural history of human papillomaviruses (HPV) and cervical neoplasia. Over a period of 18 months, ending in December 1994, 10,080 women were recruited into our study, after informed consent was obtained. At the initial recruitment visit, all women were administered a brief risk factor questionnaire, had 15ml of blood collected and, if sexually active, were given a pelvic examination. At the time of the pelvic examination, a Pap smear was collected, as were additional cervical cells which were then used for additional monolayer smears (ThinPrep) and for human papillomavirus and other testing. Pictures of the cervix, known as cervigrams, were also taken as a third screening test. Based on these screening tests, women were referred to colposcopy, at which time a more detailed risk factor questionnaire was administered, additional cervical cells and blood (15ml) were collected, and histological specimens were obtained, if indicated by the colposcopy. Women diagnosed with a high-grade cervical lesion (HSIL) or cervical cancer were treated by Social Security Administration clinicians using standard local protocols.

Women without evidence of HSIL or cancer at enrollment comprise the group of subjects who have been followed as part of our longitudinal study. Three distinct groups of women of approximately equal size (about 3,000 women each) exist within our longitudinal cohort. The first group consists of women who at enrollment had evidence of low-grade cervical lesions (LSIL) or equivocal lesions and a sample of the remaining cohort members. This group is being followed actively at 6-12 month intervals through their seventh anniversary in the cohort. The second group consists of women who were cytologically normal at enrollment but randomly selected for active follow-up. This second group will be seen once after enrollment, at their fifth anniversary in the cohort. Women in this group with evidence of LSIL at the fifth anniversary visit will be added to the first group described above and followed at 6-month intervals. The final group consists of the remaining women in our cohort (all cytologically normal at enrollment). These women are being followed passively via linkage to the cytology and tumor registries in Cost Rica.

Clinical visits conducted during follow-up consist of a brief personal interview that collects information on exposures since enrollment, the collection of 15ml blood, and a pelvic examination. Pap smear is prepared during the pelvic examination, and additional cervical specimens are collected and used to prepare a monolayer smear (ThinPrep) and for human papillomavirus and other testing. Similar to the enrollment visit, cervigrams are also collected from each participant at the time of their follow-up visits.

During follow-up, women with any evidence of progression to HSIL or cancer (by Pap smear, ThinPrep, cervicography, or by visual inspection) are referred to colposcopy, censored from the study, and treated by Social Security Administration clinicians using standard local protocols.

DETAILED DESCRIPTION:
A population-based study was initiated in Costa Rica in June 1993 to investigate the natural history of human papillomaviruses (HPV) and cervical neoplasia. Over a period of 18 months, ending in December 1994, 10,080 women were recruited into our study, after informed consent was obtained. At the initial recruitment visit, all women were administered a brief risk factor questionnaire, had 15ml of blood collected and, if sexually active, were given a pelvic examination. At the time of the pelvic examination, a Pap smear was collected, as were additional cervical cells which were then used for additional monolayer smears (ThinPrep) and for human papillomavirus and other testing. Pictures of the cervix, known as cervigrams, were also taken as a third screening test. Based on these screening tests, women were referred to colposcopy, at which time a more detailed risk factor questionnaire was administered, additional cervical cells and blood (15ml) were collected, and histological specimens were obtained, if indicated by the colposcopy. Women diagnosed with a high-grade cervical lesion (HSIL) or cervical cancers were treated by Social Security Administration clinicians using standard local protocols.

Women without evidence of HSIL or cancer at enrollment comprise the group of subjects who were followed as part of our longitudinal study. Three distinct groups of women of approximately equal size (about 3,000 women each) exist within our longitudinal cohort. The first group consists of women who at enrollment had evidence of low-grade cervical lesions (LSIL) or equivocal lesions and a sample of the remaining cohort members. This group was followed actively at 6-12 month intervals through their seventh anniversary in the cohort. The second group consists of women who were cytologically normal at enrollment but randomly selected for active follow-up. This second group was seen once after enrollment, close to fifth anniversary in the cohort. Women in this group with evidence of LSIL at the fifth anniversary visit were added to the first group described above and followed at 6-month intervals. The final group consists of the remaining women in our cohort (all cytologically normal at enrollment). These women were followed passively via linkage to the cytology and tumor registries in Costa Rica.

Clinical visits conducted during follow-up consisted of a brief personal interview that collects information on exposures since enrollment, the collection of 15ml blood, and a pelvic examination. A Pap smear was prepared during the pelvic examination, and additional cervical specimens were collected and used to prepare a monolayer smear (ThinPrep) and for human papillomavirus and other testing. Similar to the enrollment visit, cervigrams were also collected from each participant at the time of their follow-up visits.

During follow-up, women with any evidence of progression to HSIL or cancer (by Pap smear, ThinPrep, cervicography, or by visual inspection) were referred to colposcopy, censored from the study, and treated by Social Security Administration clinicians using standard local protocols.

ELIGIBILITY:
* INCLUSION CRITERIA FOR FOLLOW-UP PHASE OF NATURAL HISTORY STUDY:

Less than 35 years of age.

Intact uterus (non-hysterectomized).

In good general health.

Non-pregnant.

For women not using OCs: Having regular cycles [cycles 25-35 days in length].

HPV16 seropositive [based on data from latest visit tested].

No evidence of HSIL/cancer [based on data from latest visit within cohort].

Willing to participate [informed consent].

INCLUSION CRITERIA FOR FOLLOW-UP PHASE OF COHORT STUDY:

Must be between the ages of 45 to 70 years.

Women who do not have a final diagnosis of HSIL.

Ages: 18 Years to 100 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: A population-based study was initiated in Costa Rica in June 1993 to investigate the natural history of human papillomaviruses (HPV) and cervical neoplasia. Over a period of 18 months, ending in December 1994, 10,080 women were recruited into our study, after informed consent was obtained. Three distinct groups of women of approximately equal size (about 3,000 women each) exist within our longitudinal cohort. The first group consists of women who at enrollment had evidence of low-grade cervical lesions (LSIL) or equivocal lesions and a sample of the remaining cohort members. The second group consists of women who were cytologically normal at enrollment but randomly selected for active follow-up. The final group consists of the remaining women in our cohort (all cytologyically normal at enrollment).
Sampling Method: Probability Sample
Enrollment: 11545 (Actual)
Dates: Start 1999-05-20 (Actual); Primary Completion 2012-03-12 (Actual); Study Completion 2012-03-12 (Actual)

PRIMARY OUTCOMES:
Natural History of human papillomaviruses (HPV) and cervical neoplasia | 7-year follow-up
  Cervical precancer and cancer

CONTACTS AND LOCATIONS:
Overall Officials: Mark H Schiffman, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- Costa Rican Social Security Administration, Tres Ríos, Costa Rica

REFERENCES:
- [Background] Campos NG, Burger EA, Sy S, Sharma M, Schiffman M, Rodriguez AC, Hildesheim A, Herrero R, Kim JJ. An updated natural history model of cervical cancer: derivation of model parameters. Am J Epidemiol. 2014 Sep 1;180(5):545-55. doi: 10.1093/aje/kwu159. Epub 2014 Jul 31. PMID 25081182